CLINICAL TRIAL: NCT00091351
Title: A Phase III Randomized Study of Preoperative Radiation Plus Surgery Versus Surgery Alone for Patients With Retroperitoneal Sarcomas (RPS)
Brief Title: Surgery With or Without Radiation Therapy in Treating Patients With Primary Soft Tissue Sarcoma of the Retroperitoneum or Pelvis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z9031; ACOSOG-Z9031; CDR0000387803 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Sarcoma
Keywords: adult alveolar soft-part sarcoma; adult angiosarcoma; adult epithelioid sarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; adult malignant fibrous histiocytoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Experimental): Patients undergo surgery.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed at 28 days, 4 months, every 6 months for 5 years, and then annually for 5 years.
  Interventions: Procedure: conventional surgery
- radiation + surgery (Experimental): Patients undergo preoperative radiotherapy once daily, 5 days a week, for 5.5 weeks. Within 28-63 days after the completion of radiotherapy, patients undergo surgery.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed at 28 days, 4 months, every 6 months for 5 years, and then annually for 5 years.
  Interventions: Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: conventional surgery
Radiation: radiation therapy
  Arms: radiation + surgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy before surgery may shrink the tumor so that it can be removed. It is not yet known whether surgery is more effective with or without radiation therapy.

PURPOSE: This randomized phase III trial is studying surgery alone to see how well it works compared to radiation therapy together with surgery in treating patients with primary soft tissue sarcoma of the retroperitoneum or pelvis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with primary soft tissue sarcoma of the retroperitoneum or pelvis treated with surgery with vs without preoperative radiotherapy.

Secondary

* Compare the toxicity and complications associated with these regimens in these patients.
* Compare the rate of microscopically complete surgical resection in patients treated with these regimens.
* Compare the overall survival rate of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor grade (low [G1] vs intermediate [G2] vs high [G3/4]), tumor size (< 15 cm vs ≥ 15 cm), and tumor histology (liposarcoma vs non-liposarcoma). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo surgery.
* Arm II: Patients undergo preoperative radiotherapy once daily, 5 days a week, for 5.5 weeks. Within 28-63 days after the completion of radiotherapy, patients undergo surgery.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 28 days, 4 months, every 6 months for 5 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 370 patients (185 per treatment arm) will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary soft tissue sarcoma of the retroperitoneum or pelvis (e.g., iliac fossa)

  * The following histologies are eligible:

    * Alveolar soft part sarcoma
    * Anaplastic sarcoma
    * Angiosarcoma
    * Atypical lipomatous tumor (low-grade liposarcoma)
    * Clear cell sarcoma
    * Epithelioid sarcoma
    * Fibrosarcoma
    * Leiomyosarcoma
    * Liposarcoma (all subtypes)
    * Malignant fibrous histiocytoma
    * Malignant peripheral nerve sheath tumor
    * Myxofibrosarcoma
    * Neurofibrosarcoma
    * Spindle cell sarcoma
    * Synovial sarcoma
    * Unclassified sarcoma
  * The following histologies are not eligible:

    * Rhabdomyosarcoma
    * Extraosseous Ewing's sarcoma
    * Primitive neuroectodermal tumor
    * Osteosarcoma
    * Chondrosarcoma
    * Aggressive fibromatosis (desmoid tumor)
    * Gastrointestinal stromal tumor
    * Sarcomatoid carcinoma
    * Hemangiopericytoma
* Retroperitoneal sarcomas located predominantly in the retroperitoneum extending across the inguinal ligament into the abdominal wall are allowed provided that ≥ 90% of the tumor volume is located within the retroperitoneal space

  * No bowel obstruction OR history of previous bowel obstruction attributed to retroperitoneal tumor
* Primary non-visceral retroperitoneal masses consistent with sarcoma allowed provided diagnoses of carcinoma, melanoma, and lymphoma are excluded by immunohistochemistry
* Measurable gross disease by abdominopelvic CT scan (with IV and oral contrast) or MRI (with IV contrast)
* Patients must have undergone radiotherapy consultation within the past 30 days to confirm the feasibility of preoperative external-beam radiotherapy
* Patients must have undergone surgical consultation within the past 30 days to confirm and document the feasibility of macroscopically complete resection

  * No prior macroscopically incomplete (R2) resection (i.e., partial debulking or subtotal tumor resection with gross residual disease)
* No pelvic sarcoma extending through the sciatic notch
* No clinical or radiographic evidence of probable metastatic disease

  * Equivocal pulmonary or liver lesion allowed provided the likelihood of metastatic disease is small
* No sarcoma arising from bone or any retroperitoneal viscus (except the kidney)
* No sarcoma extending across the diaphragm into the thorax
* No recurrent retroperitoneal tumor
* No multifocal disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 2,500/mm^3
* Platelet count ≥ 80,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Albumin normal* NOTE: *Higher levels allowed

Renal

* Creatinine normal
* BUN normal
* Functional kidney confirmed by intravenous pyelogram and/or differential renal isotope scan

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other malignancy within the past 5 years (except effectively treated basal cell or squamous cell skin cancer) unless patient was curatively treated AND is at low risk for recurrence

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No concurrent chemotherapy for primary tumor

Radiotherapy

* No prior abdominal or pelvic irradiation
* No concurrent intraoperative or postoperative radiotherapy for primary tumor

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2004-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 5 years | at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pisters, MD, Study Chair — M.D. Anderson Cancer Center
Locations (59):
- United States (55):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (4):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario